CLINICAL TRIAL: NCT05089513
Title: Uterus Transplantation by Robotics and in Donor and Recipient
Brief Title: Uterus Transplantation by Robotics - Gothenburg III
Acronym: Robot2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Mats Brännström, Professor, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Robot 2
Record Dates: First submitted 2021-10-14; First posted 2021-10-22 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Absolute Uterine Factor Infertility
Keywords: uterus, infertility, transplantation, robotics
MeSH Terms: conditions — Infertility | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic surgery (Experimental): Robotic surgery in both live donor and recipient
  Interventions: Procedure: Robotic surgery

INTERVENTIONS:
Procedure: Robotic surgery — Robotoc surgery (Da Vinci) in both donor and recipient

SUMMARY:
Robotic assisted organ procurement and robotic assisted transplantation in live donor uterus transplantation

DETAILED DESCRIPTION:
Inclusion; absolute uterine factor infertility, age between 18 and 38, BMI less than 28, non-smoker

ELIGIBILITY:
Inclusion Criteria:

Uterine factor infertility, age 18-38 years, psychological stable, in steady relationship.

Exclusion Criteria:

Smoking, systemic disease, psychological instability

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Surgical success | 0-4 months
  Uterus with viability and regular menstruations

SECONDARY OUTCOMES:
Pregnancy rate | 10-48 months
  Pregnancy rate per ET

OTHER OUTCOMES:
Live birth rate per attempted and surgically succesful transplantation | 19-72 months
  Live birth rates

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Sahlgrenska, Gothenburg, None Selected
  - Sahlgrenska University Hospital, Gothenburg

IPD SHARING:
Plan to Share IPD: No
Only group dat will be published and shared after publication, in order to avoid identification of a person